CLINICAL TRIAL: NCT06471257
Title: A Randomized, Double-blind, Multicentre, Event-driven, Parallel Group, Phase III Study Evaluating the Efficacy and Safety of PT027 Compared With PT007 Administered As Needed in Symptomatic Chinese Adults With Asthma (BAIYUN)
Brief Title: A Study to Investigate Efficacy and Safety of PT027 Compared With PT007 in Symptomatic Chinese Adults With Asthma
Acronym: BAIYUN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6935C00003
Record Dates: First submitted 2024-05-29; First posted 2024-06-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Asthma; Chinese asthma population; PT027
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BDA MDI (Experimental): BDA MDI 160/180 μg (administered as 2 actuations of BDA MDI 80/90 μg)
  Interventions: Combination Product: Budesonide/Albuterol metered dose inhaler, MDI
- AS MDI (Active Comparator): AS MDI 180 μg (administered as 2 actuations of AS MDI 90 μg)
  Interventions: Combination Product: Albuterol sulfate metered dose inhaler, MDI

INTERVENTIONS:
Combination Product: Budesonide/Albuterol metered dose inhaler, MDI — Combination Product (Drug + Device)
  Other Names: PT027
  Arms: BDA MDI
Combination Product: Albuterol sulfate metered dose inhaler, MDI — Combination Product (Drug + Device)
  Other Names: PT007
  Arms: AS MDI

SUMMARY:
An event-driven, Phase III study to evaluate the efficacy and safety of BDA MDI compared with AS MDI in reducing the risk of a severe asthma exacerbation in symptomatic Chinese adults with asthma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter, event-driven, parallel group, Phase III study to assess the efficacy and safety of budesonide and albuterol metered dose inhaler (MDI) versus albuterol sulfate (AS) MDI in symptomatic Chinese adults with asthma. Both treatments will be administered as needed in response to asthma symptoms or prior to exercise. Approximately 790 participants who meet the eligibility criteria will be randomized.

The study will consist of 3 periods:

1. Screening period: 14 to 28 days
2. Treatment period: minimum of 24 weeks and maximum of 52 weeks
3. Safety follow-up period: occur 2 weeks (± 4 days) after Visit 8, EOS or PDV, whichever occurs first

790 participants who meet the eligibility criteria will be randomly assigned in a 1:1 ratio to receive one of the following 2 treatments to be used as reliever therapy on top of usual maintenance treatment:

* BDA MDI 160/180 μg (administered as 2 actuations of BDA MDI 80/90 µg) as needed
* AS MDI 180 μg (administered as 2 actuations of AS MDI 90 μg) as needed

ELIGIBILITY:
Inclusion Criteria:

1. Documented physician-diagnosed asthma for at least 12 months prior to Visit 1
2. Receiving 1 of the scheduled asthma maintenance therapies for 3 months with stable dosing for at least the last 4 weeks before Visit 1
3. Pre-bronchodilator FEV1 of ≥ 40% to < 90% predicted normal value for adults.
4. Documented reversibility to albuterol
5. A documented history of at least one severe asthma exacerbation within 12 months before Visit 1
6. ACQ-7 score ≥ 1.5 assessed at Visit 1
7. ACQ-5 score ≥ 1.5 assessed at Visit 2
8. Receiving inhaled SABA as needed prior to Visit 1 for at least 3 months
9. Use of Sponsor-provided salbutamol sulfate inhalation aerosol as needed medication due to asthma symptoms on at least 3 days during the last week of the run-in period before Visit 2
10. Demonstrate acceptable MDI administration technique as assessed by the investigator; use of spacers is prohibited
11. Able to perform acceptable and reproducible PEF measurements as assessed by the investigator
12. BMI < 40 kg/m2
13. Negative pregnancy test (urine at Visit 1) for female participants of childbearing potential
14. Women of childbearing potential must agree to prevent pregnancy
15. Compliance: must be willing to remain at the study site as required per protocol and complete all visit assessments

Exclusion Criteria:

1. Chronic obstructive pulmonary disease or other significant lung disease
2. Oral/SCS use (any dose) within 6 weeks before Visit 1
3. Chronic use of OCS ≥ 3 weeks use in 3 months prior to Visit 1
4. Having received any marketed or investigational biologic within 3 months or 5 half-lives before Visit 1, whichever is longer, or any other prohibited medication
5. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months before Visit 1
6. Life-threatening asthma as defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s) within last 5 years of Visit 1
7. Completed treatment for lower respiratory infection or asthma exacerbation within 6 weeks of Visit 1
8. Upper respiratory infection involving antibiotic treatment not resolved within 7 days before Visit 1
9. Clinically significant laboratory abnormalities
10. Historical or current evidence of a clinically significant disease
11. Cancer not in complete remission for at least 5 years before Visit 1
12. History of psychiatric disease, intellectual deficiency, poor motivation, or other conditions if their magnitude is limiting informed consent validity
13. Have a known or suspected hypersensitivity to albuterol/salbutamol, or budesonide and/or their excipients
14. Inability to abstain from protocol-defined prohibited medications during the study
15. Having received a live attenuated vaccination within 7 days of Visit 1
16. Currently pregnant or breastfeeding
17. Participants who experience > 1 asthma exacerbation during the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation | 24 to 52 weeks
  The efficacy of BDA MDI administered as needed compared with AS MDI on severe asthma exacerbation risk over the 24 to 52 week treatment period.

SECONDARY OUTCOMES:
Severe asthma exacerbation rate (annualized) | 24 to 52 weeks
  The efficacy of BDA MDI administered as needed compared with AS MDI on severe asthma exacerbations and SCS exposure
Total SCS exposure over the treatment period | 24 to 52 weeks
  The efficacy of BDA MDI administered as needed compared with AS MDI on severe asthma exacerbations and SCS exposure
ACQ-5 responder (≥ 0.5 decrease) | Week 24
  The effect of BDA MDI administered as needed compared with AS MDI on PROs at Week 24
AQLQ+12 responder (≥ 0.5 increase) | Week 24
  The effect of BDA MDI administered as needed compared with AS MDI on PROs at Week 24

CONTACTS AND LOCATIONS:
Locations (67):
- China (66):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chizhou
  - Research Site, Chongqing
  - Research Site, Dazhou
  - Research Site, Deyang
  - Research Site, Ganzhou
  - Research Site, Guangyuan
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Heifei
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Luoyang
  - Research Site, Luzhou
  - Research Site, Mianyang
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Panjin
  - Research Site, Panzhihua
  - Research Site, Pingxiang
  - Research Site, Qingdao
  - Research Site, Rui’an
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuhu
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xintai
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yibin
  - Research Site, Yinchuan
  - Research Site, Yueyang
  - Research Site, Yuhuan
  - Research Site, Zhangzhou
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
  - Research Site, Zhuji
  - Research Site, Zibo
  - Research Site, Zigong
  - Research Site, Zunyi
- Research Site, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home